CLINICAL TRIAL: NCT06752512
Title: Remote Temperature Monitoring of Patients At Risk for Developing Fever
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AION Biosystems (Industry)
Collaborators: Ellis Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ELLIS001
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Fever; Cancer; Remote Patient Monitoring
Keywords: fever; infection; sepsis; cancer; chemotherapy; immunocompromised; temperature; wearable; remote patient monitoring
MeSH Terms: conditions — Fever; Neoplasms; Infections; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Remote Patient Monitoring (Experimental): Patients assigned remote patient monitoring
  Interventions: Device: Remote Patient Monitoring

INTERVENTIONS:
Device: Remote Patient Monitoring — 24/7 remote patient monitoring with a wearable thermometer
  Other Names: RPM

SUMMARY:
The purpose of this program is to evaluate remote temperature monitoring in cancer patients at risk of fever and infection due to chemotherapy treatment. The main questions it aims to answer are:

* does remote temperature monitoring reduce the number of days spent inpatient
* what out-of-pocket cost can a patient expect to incur for participating in remote temperature monitoring
* the number of billable CPT codes that will be generated by providing remote temperature monitoring

Researchers will compare compliant and non-compliant patients to assess if compliance with remote temperature monitoring is associated with a decrease in the number of days spent inpatient.

Patients will

* wear the thermometer for the duration of their participation in the study
* have their temperature monitored continuously
* receive alerts on their phone when their temperature exceeds a threshold for a sustained duration, configurable by their physician
* respond to texts or calls from remote monitors when an alert is triggered

ELIGIBILITY:
Inclusion Criteria:

* Subject is at risk of a fever post discharge.
* Subject is ≥ 18 years or older.
* Subject has an iOS or Android phone, or is able to operate an AION provided smartphone device.
* Subject is willing to install the TempShield app on his/her phone.
* Subject is willing to allow AION to send text reminders to take temperature or complete surveys.
* Subject is willing to take an oral temperature as directed by their care plan.
* Subject is willing to configure the phone to ensure these notifications are delivered, even when phone is in a "no notification" mode.
* Subject or subject caretaker is able and willing to complete subject surveys.
* Subject is willing and able to provide written informed consent in English.
* Subject is willing and able to comply with all program procedures, requirements, assessments, visits, and complete questionnaires.
* English speakers

Exclusion Criteria:

* Unable to provide informed consent
* Subjects with a history of Medical Adhesive-Related Skin Injury (MARSI)
* Subjects with no available placement that avoids open wounds or traumatized skin (burns. Blisters. Etc.)
* Non-English speakers: The mobile application is only currently available in English. Future development will include other languages.
* Subjects receiving prophylactics that could induce fever.
* Subjects with a silicon allergy
* Subject does not have iOS or Android phone, and is unable to operate an AION provided smartphone device.
* Subjects who are not willing to take an oral temperature per their care plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Mean number of inpatient days | Day of enrollment to the end of participation in the study, a maximum of 180 days after enrollment
  The number of days the participant was admitted to a hospital while receiving remote patient monitoring

SECONDARY OUTCOMES:
Mean out-of-pocket cost | Day of enrollment
  The patient's out-of-pocket expense for setup of remote patient monitoring
Number of CPT codes generated | Day of enrollment to the end of participation in the study, a maximum of 180 days after enrollment
  Number of CPT codes generated for remote patient monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Tallat Mahmood, M.D., Principal Investigator — Ellis Hospital
Locations (1):
- Ellis Hospital, Schenectady, New York, United States

IPD SHARING:
Plan to Share IPD: No